CLINICAL TRIAL: NCT01579604
Title: Early Nerve Reconstruction Approach in Tetraplegic Patients With Dysfunctional Upper Extremity: a Randomized Controlled Trial.
Brief Title: Nerve Transfer Reconstruction in the Tetraplegic Upper Extremity
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Sean Bristol, Principal Investigator, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H11-02475
Record Dates: First submitted 2012-03-22; First posted 2012-04-18 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Tetraplegia; Plegia; Paresis; Cervical Spinal Cord Injury
Keywords: Loss of upper extremities functions; Nerve transfer
MeSH Terms: conditions — Quadriplegia; Paralysis; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgical arm (Experimental): Nerve reconstruction:
  Early nerve transfer (around 6-9 months post cervical spine injury) will be performed in this group of patients.
  Interventions: Procedure: Nerve reconstruction
- Non-surgical (or observed) (No Intervention): Patients in this group will receive standard of care and be observed for up to two years post injury.

INTERVENTIONS:
Procedure: Nerve reconstruction — Under general anesthetic, the surgeon will make a cut on the back (dorsal) part of the forearm. The radial nerve will be identified and specifically the branches which control the supinator muscle and the remainder of the radial nerve (Posterior interosseous nerve or PIN). . The PIN branch will be stimulated to ensure that it is non-functional. Then, the supinator branch will be stimulated to ensure it is functioning and is appropriate for transfer. If appropriate, the supinator branch will be severed and connected to the EDC branch under the operating room microscope. After the surgery, the patient will be placed into a splint including the forearm and hand for 2-3 weeks.
  Arms: Surgical arm

SUMMARY:
The cervical spine is most commonly injured, accounting for 53.4% of spinal injuries. More than 40% of all spinal injuries occur at either C4, C5 or C6 levels leading to variable loss of function in the upper extremities.

Traditionally, patients sustaining a cervical spine injury were followed for 2 years to ensure that recovery had stabilized before offering upper extremity reconstruction. This type of reconstruction includes active muscle transfer, tendon transfer and joint fusion.

Patients are most commonly assessed immediately at the time of injury. Muscle testing is commonly performed using Medical Research Grading System (MRC).

Although complete neurologic stabilization may not be complete until 2 years post-injury, in the group with initial grade 0 muscle strength after the acute phase of injury, expectations of improved muscle strength to or beyond grade 3 after 4-6 months is minimal. And grade 3 muscle strength is felt to be the minimum useful functional strength in a muscle group.

The investigators propose an early nerve reconstruction approach to the tetraplegic patient with dysfunction of the upper extremity to augment the available tendon transfers.

A comparative pilot study is proposed to determine the effectiveness of supinator branch to posterior interosseous nerve (PIN) transfer in 5 patients with cervical spine injury. Patient who fits inclusion criteria will be offered the opportunity to be involved in the study and reviewed at 6 months from injury. If the patient still has not regained Grade 3 power in finger or thumb extension, they will be randomized to be in a surgical group or non-surgical group.

If informed consent is obtained, then surgery will be completed between 6-9 months from the patient's original cervical spine injury. The patient will be followed at regular intervals post-operatively with expectation of 18-24 month follow-up.

Measures will be used pre and post-operatively for comparison. Measures will include MRC muscle grade (EDC), range of motion, Disability of the Arm, Shoulder, and Hand Questionnaire (DASH), and The Graded Redefined Assessment of Strength Sensibility and Prehension (GRASSP) (Kalsi-Ryan, 2011).

DETAILED DESCRIPTION:
There is currently no published data showing the effect of early nerve transfer on hand function recovery of the subset of tetraplegic patients, who have initial grade 0 muscle strength immediately after their injuries. We are interested in conducting a pilot study comparing the surgical group to the non-surgical group. A larger trial will be planned if the preliminary results show positive improvement in hand function recovery.

ELIGIBILITY:
Inclusion Criteria:

* Cervical spine injury with functional loss in the upper extremity
* Greater than 4 months out from C-spine injury
* Stable motor recovery
* Medically stable
* International Classification for Surgery of the Hand in Tetraplegia of 0-5 at 6 months
* Grade 0 finger/thumb extension at 6 months
* Subjects fluent in English or when not fluent, an appropriate translator is present

Exclusion Criteria:

* Unstable patient
* Joint contracture
* Spasticity
* Loss of function is expected to be improved by reliable tendon transfer, tenodesis or arthrodesis that is available
* Evidence of recovering finger/thumb extension at 4-6 months
* Greater than 12 months from spinal cord injury
* Subject not fluent in English or an appropriate translator not available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-06; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Medical Research Grading (MRC) System | Baseline (before surgery)
  A grading system testing the strength of muscles and ranging from grade 0 (weakest) to grade 5 (strongest).
Medical Research Grading (MRC) System | 9 months post-op
  A grading system testing the strength of muscles and ranging from grade 0 (weakest) to grade 5 (strongest).
Medical Research Grading (MRC) system | 12 months post-op
  A grading system testing the strength of muscles and ranging from grade 0 (weakest) to grade 5 (strongest).
Medical Research Grading (MRC) system | 24 months post-op
  A grading system testing the strength of muscles and ranging from grade 0 (weakest) to grade 5 (strongest).

SECONDARY OUTCOMES:
Range of motion | Baseline (before surgery)
  Measurement of distance and direction of a which a joint can move compared to its full potential.
Range of motion | 9 months post-op
  Measurement of distance and direction of a which a joint can move compared to its full potential.
Range of motion | 12 months post-op
  Measurement of distance and direction of a which a joint can move compared to its full potential.
Range of motion | 24 months post-op
  Measurement of distance and direction of a which a joint can move compared to its full potential.
DASH questionnaire | Baseline (before surgery)
  A validated instrument used as a measure of the function of upper extremity.
DASH questionnaire | 9 months post-op
  A validated instrument used as a measure of the function of upper extremity.
DASH questionnaire | 24 months post-op
  A validated instrument used as a measure of the function of upper extremity.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Bristol, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada